CLINICAL TRIAL: NCT05286307
Title: Adductor Canal Block and IPACK Block vs. Isolated Adductor Canal Block for Post-Operative Analgesia Following ACL Reconstruction With Bone Patellar Tendon Bone Autograft: A Single Center Randomized Placebo-Controlled Trial
Brief Title: Adductor Canal Block and IPACK Block vs. Isolated Adductor Canal Block for Post-Operative Analgesia Following ACL Reconstruction With Bone Patellar Tendon Bone Autograft:
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-00148
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving IPACK block (Experimental): Patients in this study group will receive the standard of care adductor canal block composed of 15 mL of Bupivacaine (0.25%). And receive the additional IPACK block performed using 20 mL of Bupivacaine (0.25%) injected into the interspace between the popliteal artery and capsule of the knee.
  Interventions: Drug: IPACK block
- Standard of care group (No Intervention): Patients in the control group will receive the standard of care adductor canal block composed of 15 mL of Bupivacaine (0.25%).

INTERVENTIONS:
Drug: IPACK block — IPACK block with 20 mL of 0.25% Bupivacaine injected into the Interspace between the Popliteal Artery and Capsule of the Knee
  Arms: Participants receiving IPACK block

SUMMARY:
A randomized, single-blind, single-center study measuring the effects of adductor canal block combined with IPACK infiltration compared to adductor canal block alone on post-operative pain and opioid consumption in patients undergoing ACL reconstruction with Bone Patellar Tendon Bone Autograft

DETAILED DESCRIPTION:
The protocol will determine if the addition of an IPACK block to the standard adductor canal block is superior to an isolated adductor canal block in controlling post-operative pain and decreasing postoperative opioid consumption in patients undergoing ACLR with Bone Patellar Tendon Bone Autograft

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age
* Patients undergoing primary ACL reconstruction with BPTB Autograft
* ASA I or II

Exclusion Criteria:

* Patients younger than 18 and older than 75.
* Patients with multi-ligament injury
* Patients undergoing concomitant cartilage procedure or osteotomy.
* Patients with a history of chronic pain that have used opioids for pain management for 3 months or longer.
* Patients who are allergic to oxycodone;
* Patients with diagnosed or self-reported cognitive dysfunction;
* Patients with a history of neurologic disorder that can interfere with pain sensation;
* Patients with a history of drug or recorded alcohol abuse;
* Patients who are unable to understand or follow instructions;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
* Patients with an allergy or contraindication to any of the medications used in the study, or patients with a contraindication to any study procedures;
* Patients with a BMI over 45;
* Any patient that the investigators feel cannot comply with all study related procedures;
* Any pregnant patient; assessed via urine pregnancy test in the preoperative area as part of standard preoperative surgical protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be maintained in an encrypted REDCap database to be accessed only by the principal investigator and study team members

REFERENCES:
- [Derived] Rao N, Triana J, Avila A, Campbell KA, Alaia MJ, Jazrawi LM, Furiguele D, Popovic J, Strauss EJ. Postoperative Pain and Opioid Usage With Combined Adductor Canal and IPACK Block Versus Isolated Adductor Canal Block After Anterior Cruciate Ligament Reconstruction With a Bone-Patellar Tendon-Bone Autograft: A Single-Center Randomized Controlled Trial. Am J Sports Med. 2025 May;53(6):1359-1367. doi: 10.1177/03635465251328609. Epub 2025 May 1. PMID 40308075

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Started | 52 | 50
Completed | 24 | 12
Not Completed | 28 | 38
Not completed — Incomplete outcome assessments | 2 | 1
Not completed — Discovery of multi-ligamentous injury intra-operatively | 0 | 1
Not completed — Lost to follow up at 6 months | 25 | 35
Not completed — Study medication not available | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.88 (7.42) | 29.67 (10.38) | 28.47 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 10 | 34
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 14 | 8 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Opioid Utilization in First 24 Hours Post-Surgery
Description: Opioid utilization for the first 24 hours after surgery, including during surgery, is calculated as oral morphine equivalent.
Time Frame: Up to Hour 24 Post-Operation
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 49 | 47
morphine milligram equivalents | 6.1 (5.5) | 10.7 (7.1)

2. Secondary Outcome: Patient-Reported Visual Analog Scale (VAS) Scores at 24 Hours Post-Surgery
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score ranges from 0 (no pain) to 100 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Hour 24 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 49 | 47
score on a scale | 55.2 (18.8) | 67.7 (26.3)

3. Secondary Outcome: Patient-Reported VAS Scores at 48 Hours Post-Surgery
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 100 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Hour 48 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 49 | 46
score on a scale | 55.5 (24.34) | 64 (22.6)

4. Secondary Outcome: Patient-Reported VAS Scores at 72 Hours Post-Surgery
Description: as for outcome 3
Time Frame: Hour 72 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 49 | 45
score on a scale | 44.4 (23.83) | 54.9 (24.18)

5. Secondary Outcome: Patient-Reported VAS Scores at Day 7 Post-Surgery
Description: as for outcome 3
Time Frame: Day 7 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 46 | 43
score on a scale | 36.3 (23.02) | 42 (24.17)

6. Secondary Outcome: Length of Stay in Post-Anesthesia Care Unit (PACU)
Description: Measured by the length of stay after surgery (minutes)
Time Frame: Up to Day 1 Post-Operation
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 49 | 47
Minutes | 131.19 (50.47) | 131.22 (37.5)

7. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score- Physical Function Short Form (KOOS-PS)
Description: The KOOS-PS is a 7-item measure of physical functional derived from the items of the Function, daily living and Function, sports and recreational activity subscales of the KOOS. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The raw score is calculated by summing the responses and ranges from 0-28. The raw score is converted to a true interval score ranging from 0-100, where higher scores indicate greater physical function.
Time Frame: Baseline, Month 6 Post-Operation Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 24 | 12
score on a scale | 4.88 (13.6) | 13.52 (14.58)

8. Secondary Outcome: Change in Kujala Scale Score
Description: Knee pain will be measured by self reported Kujala scale. The Kujala Scale is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). The total score ranges from 0 to 100; higher scores indicate lesser knee pain.
Time Frame: Baseline, Month 6 Post-Operation Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 24 | 12
score on a scale | 9.47 (14.86) | 18.75 (19.75)

9. Secondary Outcome: Change in Tegner Activity Scale (TAS) Score
Description: The TAS asks participants to indicate the highest level of activity they are able to participate in at the time of the survey. The options range from Level 10 (competitive sports on a national elite level) to Level 0 (sick leave or disability pension because of knee problems). The total score corresponds with the selected Level and ranges from 0-10; higher scores indicate higher levels of activity.
Time Frame: Baseline, Month 6 Post-Operation Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 24 | 12
score on a scale | 1.25 (1.11) | 1.92 (1.83)

10. Secondary Outcome: Change of Range of Motion (ROM) Assessment
Description: A Range of Motion (ROM) assessment is most commonly used to measure movement of the ankles, knees, hips, shoulders, elbows, wrists and fingers. Measures of knee ROM will be taken at baseline and Month 6 to assess the change in ROM over time.
Time Frame: Baseline, Month 6 Post-Operation Visit
Population: No participants had data collected/were analyzed for the purposes of this outcome measure.
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Non-systematic assessment - self reporting by participants at follow up visits
Arm/Group | Participants Receiving IPACK Block | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05286307/Prot_SAP_000.pdf